CLINICAL TRIAL: NCT07228442
Title: A Phase 2 Study of Intratumoral Administration of L19IL2/L19TNF in Locally Advanced Cutaneous Squamous Cell Carcinoma Patients Progressing on or Intolerant to Systemic Treatment
Brief Title: L19IL2/L19TNF in Patients With Cutaneous Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2TNFSCC-06/24; 2025-523231-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-07; First posted 2025-11-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Cutaneous Squamous Cell Carcinoma
Keywords: Cutaneous Squamous Cell Carcinoma; Immune Checkpoint Inhibitor; subcutaneous lesions; locally advanced; cutaneous lesions
MeSH Terms: interventions — daromun

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): the patients will receive multiple intratumoral administrations of a mixture of L19IL2 and L19TNF to all injectable cutaneous and subcutaneous lesions once weekly for up to 4 weeks.
  Interventions: Drug: L19IL2/L19TNF

INTERVENTIONS:
Drug: L19IL2/L19TNF — intratumoral administrations

SUMMARY:
Open-label, single-arm, multicenter study in patients with locally advanced, histologically confirmed Cutaneous Squamous Cell Carcinoma (LacSCC) amenable to intratumoral injection, who have progressed on or are intolerant to Immune Checkpoint Inhibitor (ICI). The primary objective of the study is to evaluate the activity of intratumoral L19IL2/L19TNF, while the secondary objective is to assess the safety and efficacy. The patients will receive multiple intratumoral administrations of combined L19IL2 and L19TNF to all injectable cutaneous and subcutaneous lesions once weekly for up to 4 weeks: for those who have a partial response or stable disease as their best response, a second 4-week course L19IL2/L19TNF of four weekly injections may be administered as per treating physician judgement. Patients will be followed for a maximum of 160 weeks after beginning of treatment.

DETAILED DESCRIPTION:
Tumor Assessment (TA) visits will be performed at Week 8 (Day 50 from the beginning of treatment), Week 12 (Day 78), and then every 8 weeks for the first year of Follow-up (FU). During second and third years of FU, TA visits will be performed every 12 Weeks. In case a response (CR, PR) or stable disease is observed, a confirmatory assessment of the tumor response will be performed 4 weeks after the TA visit, when the response was first recorded.

Confirmation of response will be assessed by histopathological analysis of specimens from the skin treated area by multiple punch biopsies. Confirmation of tumor responses will be centrally reviewed by an independent committee (Independent Central Review, ICR).

Patients will be followed for overall survival (OS) after a relapse or progression, and any further treatment given will be recorded until LPLV. Phone contact or any other documented contact with the patient will be recorded every 6 months for OS assessment from treatment start until the death of the patient, withdrawal of consent or until study completion (LPLV).

L19IL2 or L19TNF or L19IL2/L19TNF will be administered to eligible patients under the supervision of the investigator or identified sub-investigator(s). Patients will receive intratumoral administrations of L19IL2/L19TNF into injectable cutaneous, subcutaneous tumors and nodal or in transit metastasis once weekly for up to 4 weeks. On the day of each treatment visit, all tumors to be injected should be measured and recorded (using caliper/ruler for cutaneous lesions and/or ultrasound for subcutaneous lesions). The recommended volume to be injected into the tumor(s) is dependent on the size of the lesion(s). The maximum dose to be administered in a single treatment visit is: 13 MioIU L19IL2 + 0.4 mg L19TNF. It is recommended that each lesion should receive the maximum amount possible to inject due to tumor properties at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented, locally advanced cSCC.
* Patients must have at least one injectable and measurable cutaneous or subcutaneous lesion.
* Patients must have locally advanced cSCC that has progressed on or cannot tolerate ICI treatment (adjuvant or first line) as assessed by a local multidisciplinary tumor board.
* Patients with nodal, regional or in transit injectable cSCC lesions.
* Patients must be willing to provide tissue from a core or excisional biopsy of a tumor lesion at screening and for confirmation of Objective Response or Stable Disease.
* Male or female patients, age 18 - 100 years.
* ECOG Performance Status/WHO Performance Status ≤ 2.
* Hemoglobin > 10.0 g/dL.
* Platelets > 100 x 109/L.
* ALT and AST, GGT and Lipase ≤ 1.5 x the upper limit of normal (ULN).
* Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min/1.73m2 or for patients older than 65 years without albuminuria or proteinuria, creatinine clearance < 45 mL/min/1.73m2.
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v. 5.0) Grade ≤ 1 unless otherwise specified.
* Women of childbearing potential (WOCBP) must have negative pregnancy test results at screening. WOCBP must be using, from screening to three months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group and which include, for instance, progesterone-only or combined (estrogenand progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomised partner.
* Male patients with WOCBP partners must agree to use simultaneously two acceptable methods of contraception (i.e. spermicidal gel plus condom) from the screening to three months following the last study drug administration.
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Presence of concomitant malignancies, with the exception of any cancer curatively treated more than 3 years prior to study entry and of tumors with a negligible risk for metastasis or death, such as adequately treated basal cell carcinoma of the skin (surgically removed at least 4 weeks prior to study entry), ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix, early-stage asymptomatic CLL and not under active treatment (Rai 0, Binet A) will be eligible for the study.
* Radiation therapy on the tumor sites in the 4 weeks prior to study drug administration.
* Current topical or systemic chemotherapy, immunotherapy.
* Presence of visceral metastasis.
* Presence of active severe bacterial or viral infections or other severe concurrent disease/infection requiring therapy, including positive tests for human immunodeficiency virus (HIV)-1 or HIV-2 serum antibody, hepatitis B virus (HBV), or hepatitis C virus (HCV). For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV, negative serum HBV-DNA is required. For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris, inadequately treated cardiac arrhythmias and heart insufficiency (any grade, New York Heart Association (NYHA) criteria).
* Any abnormalities observed during baseline ECG investigations that are considered clinically significant by the investigator.
* Known arterial aneurysms.
* INR > 3.
* Uncontrolled hypertension.
* Known uncontrolled coagulopathy or bleeding disorder.
* Known hepatic cirrhosis or severe pre-existing hepatic impairment.
* Moderate to severe respiratory failure.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Patients have a diagnosis of immunodeficiency or are receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions and asthma/COPD is not considered an exclusion criterion.
* Known history of allergy to IL2, TNF, or other human proteins/peptides/antibodies.
* Pregnancy or breast-feeding.
* Ischemic peripheral vascular disease (Grade IIb-IV).
* Severe diabetic retinopathy.
* Recovery from major trauma including surgery within 4 weeks prior to enrollment.
* Solid organ transplant recipient or patient with iatrogenic or pathologic severe immune suppression.
* Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Patients who have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (BORR) | From enrollment up to a maximum of 160 weeks after the start of treatment
  Best Overall Response Rate (BORR) as defined by the RECIST 1.1. criteria according to an Independent Central Review (ICR).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No